CLINICAL TRIAL: NCT06372574
Title: A Phase I, Open-Label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Anti-Tumor Activity of RO7617991 in HLA-A*02-Positive Patients With Locally Advanced and/or Metastatic MAGE-A4-Positive Solid Tumors
Brief Title: A Study of RO7617991 in Patients With Locally Advanced or Metastatic MAGE-A4-Positive Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: GO44669 study has been withdrawn due to an internal Sponsor decision. The decision was not due to any safety or efficacy concerns with the study drug.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO44669
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Refractory Cancer; Recurrent Cancer; Solid Tumor, Adult
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RO7617991 Dose Escalation and Expansion (Experimental)
  Interventions: Drug: RO7617991; Drug: Tocilizumab

INTERVENTIONS:
Drug: RO7617991 — RO7617991 will be administered by intravenous (IV) infusion. Treatment will continue until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
Drug: Tocilizumab — Tocilizumab 8 mg/kg IV will be administered to patients when necessary to treat potential cytokine release syndrome (CRS), as described in the protocol.
  Other Names: Actemra®; RoActemra®; RO4877533

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics of RO7617991, and will make a preliminary assessment of the anti-tumor activity of RO7617991 in human leukocyte antigen (HLA)-A*02 eligible patients with locally advanced or metastatic melanoma-associated antigen A4 (MAGE-A4)-positive solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Body weight ≥40 kilograms
* Life expectancy of at least 12 weeks
* Confirmed eligible HLA-A*02 genotype and tumor with confirmed MAGE-A4 expression
* Histologically confirmed locally advanced or metastatic solid tumor malignancy that has relapsed or is refractory to established therapies
* Measurable disease, according to RECIST v1.1
* Adequate hematologic and end-organ function
* Resolution to Grade ≤2 of all acute, clinically significant treatment-related toxicity from prior therapy
* An archival tumor tissue specimen or fresh baseline biopsy (when archival is not available) is required

Exclusion Criteria:

* Pregnancy or breastfeeding, or intention of becoming pregnant during the study or within 3 months after the final dose of RO7617991 or tocilizumab
* Clinically significant cardiopulmonary dysfunction
* Clinically significant liver disease
* Poorly controlled Type 2 diabetes mellitus
* Active hepatitis B or C infection
* Positive test for human immunodeficiency virus (HIV)
* History of allergic reactions to red meat or tick bites or known galactose-alpha-1,3-galactose (alpha-gal) hypersensitivity
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Symptomatic pleural effusion, pericardial effusion, or ascites or any prior procedural intervention for pleural effusion, pericardial effusion, or ascites within 6 weeks prior to enrollment
* Active or history of autoimmune disease or immune deficiency
* Treatment with systemic immunosuppressive medications
* Prior allogeneic stem cell or solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | From first dose until 90 days after the final dose of study treatment (up to approximately 3 years)
Number of Participants with Abnormal Values in Targeted Vital Signs | From Baseline (predose) until 90 days after the final dose of study treatment (up to approximately 3 years)
  The targeted vital signs include pulse rate, respiratory rate, systolic and diastolic blood pressure, pulse oximetry, and body temperature.
Number of Participants with Abnormal Values in Clinical Laboratory Test Parameters | From Baseline (predose) until 90 days after the final dose of study treatment (up to approximately 3 years)

SECONDARY OUTCOMES:
Serum Concentration of RO7617991 at Specific Timepoints | From first dose until 30 days after the final dose of study treatment (up to approximately 3 years)
Objective Response Rate (ORR), as Determined by the Investigator According to RECIST v1.1 | From Baseline until until radiographic disease progression or loss of clinical benefit (up to approximately 3 years)
  RECIST v1.1 = Response Evaluation Criteria in Solid Tumors, Version 1.1
Duration of Response (DOR), as Determined by the Investigator According to RECIST v1.1 | From first occurrence of a confirmed objective response to disease progression or death, whichever occurs first (up to approximately 3 years)
Progression-Free Survival (PFS), as Determined by the Investigator According to RECIST v1.1 | From enrollment to the first occurrence of disease progression or relapse or death, whichever occurs first (up to approximately 3 years)
Overall Survival (OS) | From enrollment to death from any cause (up to approximately 3 years)
Prevalence of Anti-Drug Antibodies (ADAs) to RO7617991 at Baseline and Incidence of ADAs to RO7617991 During the Study | Baseline (predose) and from first dose until 90 days after the final dose of study treatment (up to approximately 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.

IPD SHARING:
Plan to Share IPD: No